CLINICAL TRIAL: NCT07196631
Title: A Comparison of Liposomal Bupivacaine Versus Ropivacaine for Interscalene Brachial Plexus Block in Alleviating Rebound Pain Following Shoulder Arthroscopy
Brief Title: Comparison of Liposomal Bupivacaine Versus Ropivacaine in Alleviating Rebound Pain
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Liu Jiuhong (Other)
Responsible Party: Sponsor-Investigator, Liu Jiuhong, associate professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TJMZK202507
Record Dates: First submitted 2025-09-15; First posted 2025-09-29 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Rebound Pain; Liposomal Bupivacaine
Keywords: rebound pain; Shoulder Arthroscopy; liposomal bupivacaine; ropivacaine
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: patients and outcome assessors were blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group LBP (Experimental): patients randomized to the intervention arm received 133mg of liposomal bupivacaine
  Interventions: Drug: Liposomal Bupivicaine
- group RP (Active Comparator): those in the control group received 80mg of ropivacaine
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: Liposomal Bupivicaine — patients randomized to the intervention arm received 133mg of liposomal bupivacaine
  Other Names: Ai Heng Ping
  Arms: group LBP
Drug: ropivacaine — those in the control group received 80mg of ropivacaine
  Other Names: Di Shi Li
  Arms: group RP

SUMMARY:
Shoulder arthroscopy is a frequently performed orthopedic procedure used to address various issues like rotator cuff tears, instability, and stiffness. However，postoperative pain is a common complaint, effective postoperative pain management is a crucial component to recovery after shoulder arthroscopy. For pain control after arthroscopic shoulder surgery, the interscalene brachial plexus block (IBP) is often regarded as the gold standard. It is easy to perform and has limited side effects. Nonetheless, the pain-relieving effects of the block usually last for less than 24 hours, even when using long-lasting local anesthetics like bupivacaine and ropivacaine. Considerable rebound pain is an important limitations of nerve block against postoperative pain.Its incidence is reported to be between 35% and 62% , and is more common after bone and joint surgeries, especially those involving the shoulder and knee, with a frequency 1.8 times greater than that of soft tissue operations . Therefore, it is essential to establish effective measures to avert its occurrence.Liposomal bupivacaine with its multivesicular formulation, is designed to facilitate the sustained and controlled release of bupivacaine. This formulation extended the duration of anesthetic effect and minimized rebound pain. However, studies on liposomal bupivacaine for peripheral nerve blockade have engendered great controversy. Numerous researches suggested that the use of liposomal bupivacaine for shoulder surgeries is comparable to conventional local anesthetics in terms of overall pain relief, opioids consumption, hospital stays, and postoperative complications. In this study, a randomized controlled trial with blinding of patients and outcome assessors was conducted to determine whether liposomal bupivacaine in the interscalene brachial plexus block would improve rebound pain compared to ropivacaine in patients undergoing arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
Shoulder arthroscopy represents a frequently employed orthopedic procedure for managing a wide spectrum of pathologic shoulder conditions, including rotator cuff tears, glenohumeral instability, and stiffness. Despite its minimally invasive nature, postoperative pain remains a frequent and significant concern. Effective perioperative analgesia is crucial to facilitating early mobilization and functional recovery . For this purpose, the interscalene brachial plexus block (ISBPB) remains the gold standard for postoperative pain control following arthroscopic shoulder surgery. It is easy to perform and demonstrates a favorable side effect profile. Nonetheless, the pain duration of a single-injection ISBPB is often less than 24 hours, even with long-lasting local anesthetics such as bupivacaine and ropivacaine[6]. Rebound pain following the resolution of the block poses a major challenge to the effectiveness of peripheral nerve blocks for postoperative analgesia.

Rebound pain is defined as a marked exacerbation of pain, characterized by an abrupt transition from well-controlled pain (Numerical Rating Scale, NRS ≤ 3) during the period of the block efficacy to severe pain (NRS ≥ 7) within 24 hours after peripheral nerve blockade. Reported incidence rates range from 35% to 62% , with a higher prevalence following orthopedic procedures-particularly those involving the shoulder and knee-where its frequency is 1.8 times greater compared with soft tissue operations. This rapid shift from minimal pain to intense discomfort not only disrupts sleep and impedes functional recovery, but may also negate the perioperative analgesic benefits afforded by regional anesthesia . Consequently, developing effective strategies to prevent rebound pain is critically important.

A variety of adjuncts have been evaluated to extend the duration of postoperative analgesia, with the goal of enhancing pain control and mitigating rebound pain; however, the extension of analgesia remains modest and the overall clinical benefit uncertain. While continuous peripheral nerve catheters represent an alternative means to prolong analgesia, their use is limited by technical complexity, resource intensity, and an increased risk of complications such as dislodgement or infection.

Liposomal bupivacaine, a multivesicular formulation engineered to provide sustained and controlled release of bupivacaine, has been developed to prolong analgesic duration and reduce rebound pain. Nevertheless, its efficacy in peripheral nerve blocks remains a subject of considerable debate. Multiple studies have reported that perineural administration of liposomal bupivacaine for interscalene brachial plexus block fails to significantly improve postoperative pain scores or reduce opioid consumption after shoulder surgery compared with conventional local anesthetics. Therefore, we conducted a randomized, double-blind, controlled trial to evaluate whether liposomal bupivacaine, when administered via interscalene brachial plexus block, reduces rebound pain more effectively than ropivacaine in patients undergoing arthroscopic shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* adults between 18 and 65 year-old
* American Society of Anesthesiologist (ASA) grades 1 to 3 physical classification status
* patients unilateral primary arthroscopic shoulder surgery lasting 1to 4 hours

Exclusion Criteria:

* had an allergy or intolerance to amide-type local anesthetics
* objective evidence of nerve damage in the affected upper limb
* local infection
* impaired renal function (defined as effective glomerular filtration rate < 30ml/min/1.73m2)
* coagulation disorders
* respiratory compromise（requires long term oxygen）
* had participated in another research trial involving an investigational medicinal product in the 6 months before randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
incidence of rebound pain in two groups. | up to 24 hours
  Rebound pain (RP) was defined as the abrupt transition from well-controlled pain (Numerical Rating Scale, NRS ≤ 3) during the effective period of the block to severe pain (NRS ≥ 7) within 24 hours of block performance

SECONDARY OUTCOMES:
the weighted area under the curve (AUC) for resting Numeric Rating Scale pain scores over the first 24 hours postoperatively | day 1
  the weight area under the curve (AUC) for resting Numeric Rating Scale pain scores over the first 24 hours postoperatively was accessed (Numeric Rating Scale , 0 = no pain, 10 = worst imaginable pain)
the initial onset time of pain during 72 hours | up to 72 hours
  the initial onset time of pain pain at rest was reported.
the Numeric Rating Scale pain score of initial pain happened | up to 72 hours
  the pain intensity was accessed with Numeric Rating Scale pain score (0 = no pain, 10 = worst imaginable pain)
the Numeric Rating Scale pain scores at 48 and 72 hours postoperatively | at 48 and 72 hours
  the Numeric Rating Scale pain scores at 48 and 72 hours postoperatively was accessed (0 = no pain, 10 = worst imaginable pain)
the duration of movement recovery | up to 72 hours
  the duration of movement recovery was reported as time to recovery of shoulder pendulum motion
The Numeric Rating Scale pain socre during movement | up to 72 hours
  the pain intensity during movement was accessed as shoulder pendulum motion using Numeric Rating Scale pain score (0 = no pain, 10 = worst imaginable pain)
the consumption of additional analgesics within 72 hours | up to 72 hours
  total rescue analgesic consumption within 72 hours was reported
overall patient satisfaction with pain management survey rated on a 5-point Likert scale | up to 72 hours
  overall patient satisfaction with analgesia management was rated on a 5-point Likert scale (1 = very dissatisfied, 2 = dissatisfied, 3 = unsure, 4 = satisfied, and 5 = very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Jiuhong Liu, Principal Investigator — Tongji Hospital, Tongji medical college, Huazhong University of Science and Techonology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes